CLINICAL TRIAL: NCT05414370
Title: Effects of Hyperoxia Induced Pulmonary Inflammation and Organ Injury in a Human in Vivo Model
Brief Title: Hyperoxia Induced Pulmonary Inflammation and Organ Injury: a Human in Vivo Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 18129MS-AS
Record Dates: First submitted 2022-05-11; First posted 2022-06-10 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Oxygen Toxicity; Pulmonary Injury; Acute Lung Injury
MeSH Terms: conditions — Lung Injury; Acute Lung Injury | interventions — Air

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid medical oxygen (Active Comparator): Liquid medical oxygen will be administered using high-flow nasal cannula delivery system.
  Interventions: Drug: Liquid oxygen
- Synthetic medical air (Placebo Comparator): Synthetic medical air will be administered using high-flow nasal cannula delivery system.
  Interventions: Drug: medical air

INTERVENTIONS:
Drug: Liquid oxygen — Liquid medical oxygen will be administered for 6 hours using high-flow nasal cannula delivery system with an Fi02 of 100% and flow rate of 60 litres per minute.
  Other Names: Liquid medical oxygen
  Arms: Liquid medical oxygen
Drug: medical air — Synthetic medical air will be administered for 6 hours using high-flow nasal cannula delivery system with a flow rate of 60 litres per minute.
  Other Names: Synthetic medical air
  Arms: Synthetic medical air

SUMMARY:
Oxygen is the most commonly administered therapy in critical illness. Accumulating evidence suggests that patients often achieve supra-physiological levels of oxygenation in the critical care environment. Furthermore, hyperoxia related complications following cardiac arrest, myocardial infarction and stroke have also been reported. The underlying mechanisms of hyperoxia mediated injury remain poorly understood and there are currently no human in vivo studies exploring the relationship between hyperoxia and direct pulmonary injury and inflammation as well as distant organ injury.

The current trial is a mechanistic study designed to evaluate the effects of prolonged administration of high-flow oxygen (hyperoxia) on pulmonary and systemic inflammation. The study is a randomised, double-blind, placebo-controlled trial of high-flow nasal oxygen therapy versus matching placebo (synthetic medical air). We will also incorporate a model of acute lung injury induced by inhaled endotoxin (LPS) in healthy human volunteers. Healthy volunteers will undergo bronchoalveolar lavage (BAL) at 6 hours post-intervention to enable measurement of pulmonary and systemic markers of inflammation, oxidative stress and cellular injury.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy non-smoking subjects less than 45 years of age and BMI < 29 kg/m²

Exclusion Criteria:

1. Age < 18 years
2. On concomitant medications including over the counter medications excluding oral contraception and paracetamol
3. Previous adverse reactions to LPS, lignocaine or sedative agents
4. Pregnant or Breast-Feeding
5. Participation in a clinical trial of an investigational medicinal product within 30 days
6. Consent declined
7. History of asthma or other respiratory conditions
8. Smoking/ e cigarette use
9. Marijuana use or other inhaled products with or without nicotine in the last 3 months
10. Alcohol abuse, as defined by the Alcohol Use Disorders Identification Test (AUDIT)
11. Subjects with history of prior conventional cigarette (> 100 cigarettes lifetime and smoking within 6 months) or electronic cigarette use.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Bronchoalveolar lavage Interleukin-8 (IL-8) concentration | 6 hours post-intervention
  To determine the effects of hyperoxia on alveolar inflammatory response

SECONDARY OUTCOMES:
Bronchoalveolar lavage cytokines including but not limited to tumour necrosis factor alpha, IL-1 beta and IL-6 | 6 hours post-intervention
  To determine the effects of hyperoxia on alveolar inflammatory response biomarkers
Bronchoalveolar lavage proteases and anti-proteases including but not limited to Matrix Metalloproteinases (MMP-2, MMP-8, MMP-9 and MMP-11), Tissue Inhibitors of Metalloproteinase (TIMPs 1-2) and neutrophil elastase | 6 hours post-intervention
  To determine the effects of hyperoxia on alveolar protease and antiprotease activity
Bronchoalveolar lavage white cell differential counts (total cell count, neutrophils, macrophages and lymphocytes) | 6 hours post-intervention
  To determine the effects of hyperoxia on alveolar cell populations
Plasma cytokines including but not limited to IL-8, tumour necrosis factor alpha, IL-1 beta and IL-6 | 6 and 24 hours post-intervention
  To determine the effects of hyperoxia on plasma inflammatory response biomarkers
Bronchoalveolar lavage soluble programmed cell death receptor (SP-D) | 6 hours post-intervention
  To determine the effects of hyperoxia on alveolar epithelial and endothelial function
Bronchoalveolar lavage total protein | 6 hours post-intervention
  To determine the effects of hyperoxia on alveolar epithelial and endothelial function
Bronchoalveolar lavage receptor for advanced glycation end-products (RAGE) | 6 hours post-intervention
  To determine the effects of hyperoxia on alveolar epithelial and endothelial function
Bronchoalveolar lavage 4-hydroxy-2-nonenal (4-HNE) | 6 hours post-intervention
  To determine the effects of hyperoxia on oxidative stress
Bronchoalveolar lavage oxidised low density lipoprotein (oxLDL) | 6 hours post-intervention
  To determine the effects of hyperoxia on oxidative stress
Plasma advanced glycation end products (AGE) | 6 and 24 hours post-intervention
  To determine the effects of hyperoxia on oxidative stress
Plasma oxidised low density lipoprotein (oxLDL) | 6 and 24 hours post-intervention
  To determine the effects of hyperoxia on oxidative stress
Plasma 4-hydroxy-2-nonenal (4-HNE) | 6 and 24 hours post-intervention
  To determine the effects of hyperoxia on oxidative stress

CONTACTS AND LOCATIONS:
Overall Officials: Danny McAuley, MD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Belfast Health and Social Care Trus, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Linden D, Dorrian D, Tandel S, McKelvey M, Bailey M, Conlon J, Moore D, Carr S, Taggart CC, Bradley JM, Kidney J, OKane CM, McAuley DF. Effects of Hyperoxia on Pulmonary Inflammation and organ injury in a human in vivo model (HIPI): study protocol of a randomised, double-blind, placebo-controlled trial. BMJ Open Respir Res. 2025 Feb 12;12(1):e002393. doi: 10.1136/bmjresp-2024-002393. PMID 39939102